CLINICAL TRIAL: NCT05936762
Title: Clinical Efficacy and Safety of NEOIAL HC (Hyaluronic Acid + Collagen) for Intra-articular Use in the Treatment of Severe Knee Osteoarthritis
Brief Title: Clinical Efficacy and Safety of NEOIAL HC for Intra-articular Use in the Treatment of Severe Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nextrasearch S.r.l.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoialHC
Record Dates: First submitted 2023-06-09; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis; knee; hyaluronic; collagen; neoial; gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Of the 36 screened patients, 15 had to be included and treated patients (15 as planned per-protocol). Of these, 14 patients completed the study and attended the visit at Month 6 . Since all patients were treated , the Full Analysis Set (FAS, all randomized and treated patients) was identical to the Safety Set (all treated patients).
  The mean age at enrollment was 71±7 years (range 54-80;median 73), and 12 of patients were women (85.7%) and 2 male (14.3%) . The mean BMI were26.6±3.4 (range 21-30;median 28.5) . Overall patients had knee OA with a Kellgren-Lawrence grade II and III (50/50).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoial (Experimental): Treatment with the MD
  Interventions: Device: Neoial HC

INTERVENTIONS:
Device: Neoial HC — Patients with severe knee osteoarthritis were enrolled in the clinical study and treated with 3 injections of 40 mg NEOIAL HC (HA sodium salt at 2% with two molecular weights 20% with pm at 400 kD and 80% between 1200 and 1500 kD t + collagen) at a distance of 1 week from each other, followed by a fourth infiltration of the same product at a distance of 1 month from the third.Patients were followed up with baseline clinical evaluation, reporting of adverse events after each single infiltration and subsequently at the end of treatment, 3, 6 months follow-up.

SUMMARY:
Osteoarthritis (OA) is one of the most frequent causes of pain and disability in adults. According to the Osteoarthritis Research Society International (OARSI), at least 40% of people over the age of 65 suffer from symptomatic osteoarthritis of the hip or knee. Knee osteoarthritis (OA) is the eleventh leading cause of years lived with disability according to the World Health Organization.

The guidelines show that treatment with intra-articular injections of hyaluronic acid (HA) leads to a slow, prolonged pain relief (up to six months after the first injection); On the other hand, there is little evidence in the literature about the intra-articular use of isolated collagen or in combination with hyaluronic acid in the treatment of knee osteoarthritis.

The present study showed a clinically good safety profile and provided preliminary evidence of the efficacy of NEOIAL HC for the treatment of symptomatic knee OA

ELIGIBILITY:
Inclusion Criteria:

* Age
* Knee OA
* VAS > 3
* Kellegren radiographic stage 3-4

Exclusion Criteria:

* presence of joint effusion,
* VAS score <3 according to the American College of Rheumatology Criteria
* neoplasms,
* haematological diseases,
* specific rheumatological pathologies,
* bleeding disorders, local infections,
* refusal or non-compliance of the patient,
* candidacy for knee joint replacement or any intra-articular injection during the previous year,
* addiction to opioid drugs,
* recent heart attack or stroke.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
VAS score | 6 months
  The primary objective in the study was to evaluate the mean changes from baseline at Month 3 in VAS Pain Subscale Score

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 months
  The KOOS is self-administered and assesses 5 domains: pain, symptoms, activities of daily living (ADL), sport and recreation function, and knee-related quality of life. This scale is used to evaluate knee function in terms of activities of daily living (ADL).
Lequesne | 6 months
  measure the severity for osteoarthritis for the knee (ISK). This can be used to assess the effectiveness of therapeutic interventions
Western Ontario McMaster Universities (WOMAC®) VA3.1 | 6 months
  self-administered, patient-centered health status questionnaires allowing a thorough evaluation of pain, stiffness, and knee function (24 questions through three subscales)

OTHER OUTCOMES:
occurrence of AEs and serious adverse events (SAEs) | through study completion, an average of 1 year
  reported on patients' open questionnaires, related or not to the product or procedures, abnormal laboratory results in terms of hematology, serum chemistry, and coagulation parameters, and clinically relevant findings at physical examination (including vital signs) during the entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Buda, Prof, Principal Investigator — Ospedale Santa Annunziata di Chieti
Locations (1):
- Ospedale SS Annunziata, Chieti, Italy

IPD SHARING:
Plan to Share IPD: Yes